CLINICAL TRIAL: NCT01015872
Title: The Investigation of the Roles of Prostanoids in Patients With Sleep Apnea Syndrome
Brief Title: The Roles of Prostanoids in Patients With Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Toru Oga, Respiratory Care and Sleep Control Medicine, Kyoto University, Graduate School of Medicine, Kyoto University, Graduate School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C368-kyoto
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Sleep Apnea
Keywords: sleep apnea syndrome; CPAP; prostanoids
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPAP (Experimental): the subjects introduced with CPAP treatment
  Interventions: Device: CPAP treatment

INTERVENTIONS:
Device: CPAP treatment — CPAP treatment is to improve airway obstruct for obstructive sleep apnea, and after 3 months' treatment, we evaluate the effects.

SUMMARY:
The purpose of this study is to evaluate the relationships between prostanoids and various outcomes such as sleep disturbance, hypertension and arteriosclerosis in patients with sleep apnea syndrome(SAS). In the patients introduced to continuous positive airway pressure(CPAP) treatment, the effects of CPAP are also evaluated.

DETAILED DESCRIPTION:
SAS is characterized by abnormality during sleep and hypoxemia from apnea and hypopnea, followed by systemic inflammation and organ dysfunction like cardiovascular diseases. Systemic inflammation causes the activation of arachidonic acid metabolism, producing prostaglandins (PGs) and leukotrienes (LTs). In addition, significant relationships between PGD2 and PGE2 and sleep, PGF2α and hypertension, PGI2 and thromboxane and platelet aggregation and so on are reported. Therefore, it is hypothesized that many prostanoids affect the pathophysiology of SAS. However, the relationships between prostanoids and clinical outcomes in patients with SAS are unknown. Although CPAP is the major treatment of SAS, the effects of CPAP on prostanoids are not known, either. Thus, the purpose of this study is to evaluate those relationships.

ELIGIBILITY:
Inclusion Criteria:

* Subjects hospitalized in Kyoto University Hospital for careful examination of SAS

Exclusion Criteria:

* Subjects with severe respiratory diseases, severe heart diseases, severe vascular diseases, or severe diabetes mellitus.
* Subjects taking nonsteroidal anti-inflammatory drugs, steroids or immunosuppressants.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
metabolites of arachidonic acid in the urine and blood | 3 months

SECONDARY OUTCOMES:
Polysomnography measurements | 3 months
Sleepiness and health-related quality of life | 3 months
Blood pressure and pulse rate | 3 months
Endothelial dysfunction | 3 months
Platelet aggregation | 3 months
Cardiac and neck echo cardiography | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kazuo Chin, MD, PhD, Principal Investigator — Kyoto Universuty, Graduate School of Medicine; Toru Oga, MD, PhD, Principal Investigator — Kyoto University, Graduate School of Medicine
Locations (1):
- Kyoto University, Graduate School of Medicine, Kyoto, Kyoto, Japan